CLINICAL TRIAL: NCT05514678
Title: The Effect of Cognitive Stimulation Therapy on Daily Life Activities, Depression and Life Satisfaction in Individuals With Dementia Nursing Home
Brief Title: Cognitive Stimulation Therapy for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ejdane Coskun (Other)
Responsible Party: Sponsor-Investigator, Ejdane Coskun, Lecturer, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CST in DEMENTIA
Record Dates: First submitted 2022-08-11; First posted 2022-08-24 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Dementia
Keywords: Cognitive stimulation therapy; dementia; activities of daily living; depression; life satisfaction
MeSH Terms: conditions — Dementia; Depression; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Stimulation Therapy (Experimental): In the 2nd, 3rd, 4th, 6th, 7th and 8th weeks, IPT implementation twice a week, as two themes, for 7 weeks, with each session of 45 minutes.
  Interventions: Behavioral: Cognitive Stimulation Therapy
- CST nonpharmacological intervention (Experimental): Individuals in the control group will be given two sessions in the 2nd week, and they will continue their daily lives in the following weeks.
  Interventions: Behavioral: Cognitive Stimulation Therapy

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy — CST consists of 14 sessions, each session with different themes. The materials used in therapy will differ according to the characteristics of each theme. For example; In the theme of physical games, one of the individuals will be selected by voting, and each individual will be asked to choose a song suitable for the theme and introduce himself/herself to the music accompaniment. Then, a small table game will be prepared with the rackets and ball used for table tennis, and individuals will be able to play a round of table tennis with the researcher and their groupmates. Sessions 10 min. introductory part, 25 min. activity section and 10 min. 45 minutes in total, including the ending. in progress.

SUMMARY:
Aim:

The aim of this study is to reveal the effectiveness of cognitive stimulation therapy on activities of daily living, depression and life satisfaction in individuals with mild dementia living in nursing homes.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted between 30 March-27 May 2022, with a total of 60 individuals (30 in control and 30 in intervention group) living in Adana and Seyhan Nursing Home Elderly Care and Rehabilitation Centers. The data of the study were collected with the Personal Information Form based on the literature, the Standardized Mini Mental Test (SMMT), the Barthel Activities of Daily Living Index, the Lawton and Brody Instrumental Activities of Daily Living (IADL) Scale, the Cornell Dementia in Dementia Scale (CDS) and the Satisfaction with Life Scale. In order to conduct the study, the approval of the Clinical Research Ethics Committee, written institutional permission and written permission from the participants were obtained. The individuals in the intervention group started with the introduction and pre-test application in the first week and applied CST for 45 minutes twice a week for the next 7 weeks, while the individuals in the control group started with the introduction and pre-test application in the first week and performed two sessions for one week and two days and continued their daily lives in the following weeks. The study was terminated in 9 weeks by applying the post-test to both groups in the last week. Due to the 3-month follow-up study, measurements will be made for the last time in September with the SMMT, BADL, IADL, CDS and LDL measurement tools.After being informed about the study, all individuals with dementia were given written informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with dementia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM V) by a physician
* Agree to participate in the study
* Being literate and speaking Turkish fluently
* Have communication and understanding skills
* Standardized Mini Mental Test result being between 18-23 points
* Having adequate vision and hearing functions for group participation

Exclusion Criteria:

* Presence of any sensory impairment
* Having a physical health problem that may impair group cohesion and integrity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The change of the effect of cognitive stimulation therapy on activities of daily living in individuals in nursing homes with dementia is being assessed. | up to 9 weeks
  Barthel index scores range from 0 to 100, 0-20 points; completely addicted, 21 - 61 points; severe addiction, 62 - 90 points; moderate addiction, 91 - 99 points; mild addiction, 100 points; explains independence. In studies using the Barthel Index, a score of 60 was taken as the limit, and scores above 60 explain the ability to function independently. Lawton and Brody Instrumental Daıly Lıfe Actıvıtıes Scale, the scale consists of 8 items and a single sub-dimension. The total score obtained from the scale varies between 0-8. A low score indicates a high level of addiction.
The change of the effect of cognitive stimulation therapy on depression in individuals in nursing homes with dementia is being assessed. | up to 9 weeks
  Cornell Dementia for Dementia In this scale, mood-related findings, behavioral changes, physical findings, cyclical functions and intellectual changes are evaluated with 19 items collected in 5 subgroups. Each item is scored between 0-2. A total score of eight and above suggests significant depression.
The change of the effect of cognitive stimulation therapy on life satisfaction in individuals in nursing homes with dementia is being assessed. | up to 9 weeks
  In the Satisfaction with Life Scale, a seven-point Likert type scale is graded between "strongly disagree" (1) and "strongly agree" (7). A high score on the scale indicates high life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ejdane Coşkun, Lect., Principal Investigator — ejdanecoskun@osmaniye.edu.tr
Locations (1):
- Korkut Ata University, Osmaniye, Center, Turkey (Türkiye)

REFERENCES:
- [Background] Cheng ST. Cognitive Reserve and the Prevention of Dementia: the Role of Physical and Cognitive Activities. Curr Psychiatry Rep. 2016 Sep;18(9):85. doi: 10.1007/s11920-016-0721-2. PMID 27481112
- [Background] Kurz A. [Psychosocial interventions in dementia]. Nervenarzt. 2013 Jan;84(1):93-103; quiz 104-5. doi: 10.1007/s00115-012-3655-x. German. PMID 23306213
- [Background] Aslan M, Hocaoğlu C. Psychiatric Problems Associated with Aging and Aging. Duzce University Journal of Health Sciences Institute. 2017);7(1):53-62.
- [Background] Saragih ID, Tonapa SI, Saragih IS, Lee BO. Effects of cognitive stimulation therapy for people with dementia: A systematic review and meta-analysis of randomized controlled studies. Int J Nurs Stud. 2022 Apr;128:104181. doi: 10.1016/j.ijnurstu.2022.104181. Epub 2022 Jan 22. PMID 35149325
- [Background] Aguirre E, Hoare Z, Streater A, Spector A, Woods B, Hoe J, Orrell M. Cognitive stimulation therapy (CST) for people with dementia--who benefits most? Int J Geriatr Psychiatry. 2013 Mar;28(3):284-90. doi: 10.1002/gps.3823. Epub 2012 May 10. PMID 22573599
- [Background] Aguirre E, Woods RT, Spector A, Orrell M. Cognitive stimulation for dementia: a systematic review of the evidence of effectiveness from randomised controlled trials. Ageing Res Rev. 2013 Jan;12(1):253-62. doi: 10.1016/j.arr.2012.07.001. Epub 2012 Aug 7. PMID 22889599
- [Background] Rai H, Yates L, Orrell M. Cognitive Stimulation Therapy for Dementia. Clin Geriatr Med. 2018 Nov;34(4):653-665. doi: 10.1016/j.cger.2018.06.010. Epub 2018 Aug 20. PMID 30336993
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Lok N, Buldukoglu K, Barcin E. Effects of the cognitive stimulation therapy based on Roy's adaptation model on Alzheimer's patients' cognitive functions, coping-adaptation skills, and quality of life: A randomized controlled trial. Perspect Psychiatr Care. 2020 Jul;56(3):581-592. doi: 10.1111/ppc.12472. Epub 2020 Jan 12. PMID 31930518
- See also: alzheimer's association — http://www.alzheimerdernegi.org.tr/
- See also: TUİK — https://www.tuik.gov.tr/
- See also: WHO — https://www.who.int/
- See also: WHO DEMENTİA — https://www.who.int/news-room/fact-sheets/detail/dementia